CLINICAL TRIAL: NCT07309575
Title: Regional Versus General Anesthesia for Hip Fracture and Postoperative Oxygenation
Acronym: REGENERATION
Status: Recruiting | Type: Observational
Sponsor: University of Lisbon (Other)
Collaborators: Northern Lisbon Hospital Center (Other)
Responsible Party: Principal Investigator, ANDRE DOS SANTOS ROCHA, Prof. MD PhD, University of Lisbon
Other Study IDs: CE-CAML 221/25
Record Dates: First submitted 2025-11-27; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Hip-fracture; General Anaesthesia; Regional Anaesthesia
Keywords: anaesthesia; hip femur fracture; postoperative pulmonary complications; oxygenation; sleep apnea
MeSH Terms: conditions — Hip Fractures; Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- General anaesthesia: Hip fracture surgery under general anaesthesia
- Rregional anaesthesia: Hip fracture surgery under regional anaesthesia

SUMMARY:
With this study, the investigators intend to measure oxygen saturation before and after hip surgery in the context of proximal femur fracture, comparing two types of anesthesia (general or spinal). The investigators also intend to study the effects of the two anesthetic techniques on sleep apnea, delirium, respiratory complications, and length of hospital stay.

This is an observational study, in which oxygen is measured at the fingertip with a sensor and a bracelet, without any intervention, inconvenience, or discomfort for the participant. Data will be collected on: respiratory complications, sleep apnea, delirium, length of hospital stay, and survival.

Data will be collected in the operating room and wards of Santa Maria Hospital, Lisbon, Portugal over a period of approximately 24 hours after the participant's operation. Information about participant's health and co-morbidities will be recorded.

There will be no implication for the participants' clinical care, since the study measurements will not be sent to the health professionals in charge. The operation, recovery, and treatments will not be influenced at any time by participation in the study.

DETAILED DESCRIPTION:
Frailty, comorbidities, medication (anticoagulants and anti-platellet agents) as well as acute and chronic illnesses have an impact on the choice of anesthesia strategy for hip fracture surgery. The choice between general anesthesia (GA) and loco-regional, spinal anesthesia (SA) may have impact on the postoperative period. Despite previous retrospective studies on this topic, it remains uncertain that either is superior in terms of post-operative outcomes, including mortality, delirium and respiratory complications, with conflicting results in the literature.

Postoperative pulmonary complications (PPC) are amongst the commonest complications in geriatric hip fractures, reported to be around 12%. The elder population at Hospital de Santa Maria (Tertiary University Hospital Center) receives the most challenging cases, with pilot data from the past 3 years (2022-2024, n=927) revealing an average risk score for PPC of 32,1%.

Considering that low oxygen saturation is an independent risk factor and a strong predictor for PPC, the investigators seek to compare the oxygenation during the perioperative period between the different anesthesia regimens.

The study hypothesis is that the anesthesia regimen (GA vs SA) has an impact on the oxygenation index during the first 24 postoperative hours.

The secondary objectives are to compare the sleep apnea index between GA and SA, the incidence of PPC, delirium, mortality and the length of stay (LOS) in the PACU and until discharge from the hospital.

ELIGIBILITY:
Inclusion Criteria:

* hospital admission for hip fracture;
* scheduled for hip fracture surgery;
* age above 65 years, both genders;
* capable of consent or consent by responsible person;

Exclusion Criteria:

* hip fracture during hospitalization (not present upon admission)
* patient refusal to participate

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elder subjects with hip-fracture submitted to surgery.
Sampling Method: Probability Sample
Enrollment: 102 (Estimated)
Dates: Start 2025-11-27 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Oxygenation index (SpO2/FiO2 ratio) | first postoperative day
  Oxygenation index (SpO2/FiO2 ratio) measured as the difference between oxygenation index on admission to the operating room and the mean SpO2 during the next 24 postoperative hours, compared between groups.
  Peripheral oxygen saturation measured continuously during the first postoperative day with the Konica Minolta PULSOX-DS5® device.

SECONDARY OUTCOMES:
Sleep Apnea index | first postoperative day
  average dips of SpO2 per hour, (>= 4%)
Length of stay in the Post-anestesia Care Unit | after the surgery, at discharge from the Post-anestesia Care Unit
  Length of stay in the Post-anestesia Care Unit
Hospital Length of Stay (Days) | from hospital admission to hospital discharge, approximatelly 5 days
  Length of stay in the hospital from admission until discharge, in days
postoperative pulmonary complications | during the first postoperative day
  postoperative pulmonary complications defined as hypoxemia, respiratory failure, atelectasis, pneumothorax, respiratory infection.
Delirium | during the first postoperative day
  Presence of delirium in the first postoperative day
in-Hospital mortality | From hospital admission to hospital discharge (or death), up to 3 months
  death from any cause during hospital stay, from hospital admission to discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Northern Lisbon Hospital Center, Lisbon, Lisbon District, Portugal

IPD SHARING:
Plan to Share IPD: No
only anonymised data can be shared after publication and upon reasonable request